CLINICAL TRIAL: NCT01472523
Title: A Safer Pre-Natal Diagnosis Using Free DNA in Maternal Blood
Acronym: IONA
Status: Completed | Type: Observational
Sponsor: Premaitha Health (Industry)
Responsible Party: Sponsor
Other Study IDs: 07H0607101
Record Dates: First submitted 2011-10-11; First posted 2011-11-16 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Aneuploidy, NIPT
MeSH Terms: conditions — Aneuploidy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Maternal peripheral blood samples taken in EDTA with that required for existing analysis.
  Approx 1ml of fluid from amniocentesis/chorionic villus sampling is taken additional. Patients will be followed up for 1 year after sample taken.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Controls
- Aneuploidy: T13, 18, 21 and other chromosomal abnormalities yet to be determined

SUMMARY:
A diagnostic peripheral maternal blood test taken and the free foetal DNA is analysed and the presence of trisomies using a novel method.

DETAILED DESCRIPTION:
A total of ~2000 participants have donated blood samples used for the development and validation of the IONA non-invasive prenatal screening test for Downs, Edwards and Patau syndrome. The IONA Test was CE marked Feb 2013. We are now recruiting a further 800 participants to provide blood samples to further develop and verify the test for other chromosomal abnormalities and to improve test efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Patient/subject is willing and able to give informed consent for participation in the study.
* Female, aged 16 years or above.
* Currently pregnant at time of entry to the study.
* Pregnancy having been identified as 'high-risk' by screening test.

Exclusion Criteria:

* The patient/subject may not enter the study if ANY of the following apply:
* The participant herself has Down's Syndrome or other chromosomal abnormality.
* Children under 16
* Adults with learning disabilities
* Adults who are unconscious or very severely ill
* Adults who have a terminal illness
* Adults in emergency situations
* Adults suffering from a mental illness
* Adults with dementia
* Prisoners
* Young offenders
* Adults who are unable to consent for themselves
* Any person considered to have a particularly dependent relationship with investigators

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Mothers attending clinic for routine screening. Followed up at around 1 years duration.
Sampling Method: Probability Sample
Enrollment: 1632 (Estimated)
Dates: Start 2007-04; Primary Completion 2018-02 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Validation of method of novel analysis for Aneuploidy | 2013 Approx
  Analysis of maternal blood by a selective amplification of fetal DNA over maternal DNA within that sample. Patients to be followed up for 1 year.

SECONDARY OUTCOMES:
Optimization of existing methods for maximising ffDNA | up to July 2019
  Use of novel methods either in conjugation with existing methods or as a substitute for steps in existing methodologies- currently undergoing laboratory development that could increase the titre of fetal DNA within a given sample. Patients will be followed up for 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Kelly, MBBS, Principal Investigator — National Health Service, United Kingdom
Locations (1):
- Premaitha Health, Manchester, United Kingdom